CLINICAL TRIAL: NCT02560038
Title: Phase II Trial of Paclitaxel Plus Gemcitabine and Cisplatin in Urothelial Cancer
Brief Title: Trial of Paclitaxel Plus Gemcitabine and Cisplatin in Bladder Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow enrollment; resource re-allocation
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Robert J Amato, Director and Professor, Department of Internal Medicine, Division of Oncology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-13-102; HSC-MS-13-0864 (Other: UTHealth Committee for Protection of Human Subjects)
Record Dates: First submitted 2015-09-17; First posted 2015-09-25 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Urothelial Cancer; Bladder Cancer; Metastatic
MeSH Terms: conditions — Urinary Bladder Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination chemotherapy (Experimental): Combination chemotherapy consisting of gemcitabine and cisplatin plus paclitaxel on a 21-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 will be administered as an IV infusion over 10 mg/minute on Days 1 and 8 of each cycle (each cycle is 21 days).
  Other Names: Gemzar
Drug: Paclitaxel — 175 mg/m2 will be administered as an IVPB over 3 hours on Day 2 of each cycle (each cycle is 21 days).
  Other Names: Taxol
Drug: Cisplatin — 70 mg/m2 will be administered as an IVPB over 2 hours on Day 2 of each cycle (each cycle is 21 days).
  Other Names: Platinol

SUMMARY:
This trial is for people with bladder cancer that has spread. The purpose of this research study is to see if the chemotherapy combination of gemcitabine and cisplatin plus paclitaxel is safe and effective treatment for bladder cancer.

Paclitaxel, gemcitabine and cisplatin have all been approved by the United States Food and Drug Administration (FDA). Gemcitabine and cisplatin is a standard treatment for bladder cancer. There have been studies that show that paclitaxel and cisplatin have antitumor activity in bladder cancer. European researchers studied paclitaxel, gemcitabine and cisplatin (same drug combination in this trial) and found that the combination provided good disease control and was well tolerated. Investigators are studying the same drug combination, but at different dosages and schedule.

DETAILED DESCRIPTION:
The rationale of the present study is to develop a combination based on the pharmacokinetics and mechanisms of action of the agents paclitaxel plus gemcitabine and cisplatin, which are all known active agents in urothelial tumors. Gemcitabine may be synergistic with DNA-damaging drugs such as paclitaxel and cisplatin because it can antagonize DNA repair. Investigators will investigate the combination in this Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologic demonstration of metastatic or locally unresectable transitional cell carcinoma of the urothelium. Minor components (<50% overall) of variants such as glandular or squamous differentiation, or evolution to more aggressive phenotypes, such as sarcomatoid, or small cell changes are acceptable. However, when these atypical histologies are dominant, other treatment approaches may be more appropriate, and such patients are not eligible.
* All patients must have measurable or evaluable disease. In general, liver and lung lesions should be at least 1 cm, and patients with node-only disease should have lesions of ≥ 1.5 cm in the largest dimension. Patients with disease confined to bone may be eligible if a measurable lytic defect is present. Patients with a 3-dimensional mass or pelvic sidewall fixation on bladder examination under anesthesia are considered to have measurable disease.
* All patients must have adequate physiologic reserves as evidenced by:
* Life expectancy of at least 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤2.
* No clinical history of heart disease and a normal EKG or an ejection fraction measured by echocardiogram or MUGA scan of at least 45%.
* Transaminase less than twice the upper limit of normal. Bilirubin <1.5 mg%.
* Serum creatinine ≤2.0 mg/dL. Patients presenting with obstructive uropathy may be eligible if they show excellent response to nephrostomy drainage.
* Absolute neutrophil count ≥1500; platelet count ≥100,000.
* Patients must not have had any previous systemic chemotherapy for bladder cancer, including neoadjuvant or adjuvant treatment given remotely. Gemcitabine/cisplatin is the standard of care for metastatic urothelial cancer. Patients who have received treatment would be either resistant or refractory to additional doses. In addition, they would have residual adverse effects from treatment and would be particularly susceptible to further neuropathic adverse events. Any prior intravesicular therapy is allowed.
* Women of childbearing potential must have a negative pregnancy test prior to starting therapy. Men and women of childbearing potential must be willing to consent using effective contraceptive while on treatment and for a reasonable period thereafter.
* Patients must not have an active, or likely to become active, second malignancy.
* Patients must be at least 6 weeks out from pelvic irradiation, and must not have had more than 10% of the bone marrow irradiated.

Exclusion Criteria:

* Patients with uncontrolled CNS metastasis are not eligible.
* Patients with a history of peripheral neuropathy greater than grade 1 are not eligible.
* Pregnant women are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-10; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UTHealth Memorial Hermann Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Chemotherapy
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 65 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1
  White | 1
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) Performance Status scale measures level of functioning. The scale ranges from 0 to 5, with 0 indicating the highest level of functioning and 5 the lowest.
  Participants
    ECOG score of 0 | 2
    ECOG score of 1 | 1
    ECOG score of 2 | 0
    ECOG score of 3 | 0
    ECOG score of 4 | 0
    ECOG score of 5 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy as Measured by the Objective Response Rate (ORR).
Description: Objective Response Rate (ORR) is defined as the proportion of patients achieving either a complete response or a partial response based on imaging at any time during the study. Complete response or partial response is based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Safety of Drug Regimen as Measured by Number of Adverse Events
Description: Toxicity assessment will be observational. Numbers and types of events will be quantified and graded according to CTCAE.
Time Frame: as for outcome 1
Measure: Number; unit: adverse event
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 3
adverse event | 124

3. Secondary Outcome: Efficacy as Measured by Number Who Progressed
Description: Progression is defined using RECIST 1.1 criteria: " At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)."
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: From the time the participant signs the informed consent until the participant was taken off-study or the study was stopped, an average of 6 months
Arm/Group | Combination Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Combination Chemotherapy (N=3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Fever (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomitting (Gastrointestinal disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
White Blood Cell Count Decreased (Investigations) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Perineal Pain (Reproductive system and breast disorders) | 1 (1)
Vaginal Discharge (Reproductive system and breast disorders) | 1/1 (1)
Vaginal Pain (Reproductive system and breast disorders) | 1/1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Chemotherapy (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (5)
Blood and lymphatic system disorders, Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Cardiac disorders, Swelling in center of chest around sternum (Cardiac disorders) | 1 (1)
General disorders and administration site conditions, Pretibial edema (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 1 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (7)
Rectal Fistula (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders, Thrush (Gastrointestinal disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (4)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Injury, poisoning and procedural complications, Bruise on hip (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline Phosphate increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Investigations, Elevated BUN (Investigations) | 1 (2)
Creatinine increased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (2)
Weight gain (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4)
Anorexia (Metabolism and nutrition disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder, Achiness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Vasovagal Reaction (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders, Acute renal injury (Renal and urinary disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Blood and lymphatic system disorders, Nose Bleed (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders, Angio edema (Cardiac disorders) | 1 (1)
Gastrointestinal disorders, Swollen tongue (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders, Little urine output (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination of study leading to small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT02560038/Prot_SAP_000.pdf